CLINICAL TRIAL: NCT06865183
Title: Further Evaluation of Selected Child Triple P As a Universal Intervention Delivered Through Telehealth
Brief Title: Investigating a Brief Virtual Seminar Series for Parents of Children Ages 2-12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, John Cooley, Assistant Professor, University of Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-1035c
Record Dates: First submitted 2025-02-06; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Positive Parenting Skills
Keywords: Selected Child Triple P; Parenting Intervention; Telehealth; Positive Parenting

STUDY DESIGN:
Intervention Model Description: Three study conditions compared: intervention-as-usual, intervention without an active discussion component, and waitlist control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention-as-usual (Experimental): 90-minute positive parenting seminars with active discussion component
  Interventions: Behavioral: Positive Parenting Seminar Series
- Intervention without an active discussion component (Experimental): 60-minute positive parenting seminars without an active discussion component
  Interventions: Behavioral: Positive Parenting Seminar Series
- Waitlist Control (No Intervention): Assessment-only waitlist control condition

INTERVENTIONS:
Behavioral: Positive Parenting Seminar Series — Selected Child Triple P Positive Parenting Seminar Series Delivered Through Telehealth
  Other Names: Selected Child Triple P
  Arms: Intervention without an active discussion component; Intervention-as-usual

SUMMARY:
The goal of this clinical trial is to determine whether a brief positive parenting seminar series delivered virtually helps teach parents additional tools and strategies to support healthy child development, encourage good behavior, and manage misbehavior, while improving parenting practices and child outcomes for parents of children ages 2-12.

The main questions it aims to answer are whether parents are satisfied with the intervention and find the strategies helpful and acceptable, whether the intervention leads to changes in parenting behaviors (e.g., positive parenting) and child outcomes (e.g., emotional and behavioral problems), and how removing the active discussion from the seminars impacts parents' ability to improve their parenting skills and their child's outcomes.

Researchers will compare three groups: parents receiving the seminars with a group discussion, parents receiving the seminars without a group discussion, and parents on a waitlist. This will help determine if group discussions lead to greater improvements in parenting practices and child outcomes.

Participants attended three online parenting seminars via telehealth (if assigned to a seminar group). They completed surveys before, during, and after the seminars to share their experiences and provide feedback. Participants in the waitlist group completed surveys at the beginning and end of the study, and will participate in the seminars after the study period.

DETAILED DESCRIPTION:
Despite the effectiveness of parenting interventions in promoting adaptive child-rearing behaviors and preventing youth internalizing and externalizing problems, our current model for mental health treatment that involves a highly trained mental health professional providing services in a one-on-one format at a clinic, private office, or health-care facility is not sustainable. As such, there is an urgent need to identify ways to increase the accessibility and scalability of mental health services to reduce the well-documented gap between children and families who need mental health services and those who are able to access them. Therefore, the goal of the current randomized controlled trial is to investigate the feasibility, acceptability, and preliminary efficacy of a brief (i.e., 3 session) seminar series for parents with children between the ages of 2 and 12, which was offered via telehealth to increase accessibility. Additionally, this project will evaluate whether the ability for parents to ask questions and discuss skill implementation with a mental health provider is necessary for treatment effectiveness, given that programs that do not require a provider for implementation have the potential for greater scalability.

After completing the baseline survey, eligible parents were randomly assigned to condition using block randomization. For parents assigned to the intervention-as-usual condition (i.e., 90-minute condition), seminars were delivered live by two masters-level therapists who were fully accredited in Selected Child Triple P. The seminars consisted of 60-minutes of seminar content (i.e., discussion of various parenting strategies), followed by a 30-minute question-and-answer period. Participation was encouraged by co-leaders throughout the seminars and the question-and-answer period.

For parents assigned to the intervention without an active discussion component (i.e., 60-minute condition), seminar content was pre-recorded by the same two co-leaders who led the seminars live to ensure standardization of the material and to create an environment focused on receiving information rather than active participation. During these meetings, participants were not allowed to unmute and were only able to message the hosts of the meeting (i.e., the leader).

The same seminar content was covered in both intervention conditions. The seminars included the Power of Positive Parenting, Raising Confident, Competent Children, and Raising Resilient Children.

Approximately 2-months and 4-months after attending the final seminar, parents were contacted to complete a 30-minute follow-up survey for which they were compensated. The dates that parents attended each seminar were recorded and parents were contacted approximately 2-months and 4-months after their last attended seminar (or their last opportunity to attend a seminar if they did not attend all three seminars). Parents in the waitlist control condition were contacted approximately 2-months and 4-months after the last seminar was offered to those assigned to the intervention conditions in their enrollment cohort.

ELIGIBILITY:
Inclusion Criteria:

* Parent must reside in the State of Texas
* Parent had to have at least one child ages 2-12 years
* Child had to live with parent at least one night every 2 weeks

Exclusion Criteria:

* Parent did not have sufficient English proficiency to understand seminar content and complete study-related surveys
* Parent did not have access to the internet and/or could not attend seminars using the Zoom platform
* Child was currently participating in mental health services
* Child began taking psychiatric medication within 1 month of the study
* Parent was currently participating in mental health services

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Parent Satisfaction | Weekly, through intervention completion, average of 3 weeks.
  Parents assigned to an intervention condition completed a modified 8-item version of the Parent Satisfaction Survey after each seminar. Response options ranged from 1 (Poor, No definitely not, or Not at all) to 7 (Excellent, Yes, definitely, or Very much).
Acceptability | Weekly, through intervention completion, average of 3 weeks.
  Parents assigned to an intervention condition completed a modified 9-item version of the Treatment Acceptability Rating Form. Response options ranged from 1 (Not at all) to 7 (Very much).
Positive Parenting | Baseline, 2-month, and 4-month follow-up assessments.
  All parents completed the 16-item positive parenting composite measure of the Multidimensional Assessment of Parenting Scale, which was comprised of proactive parenting (6-items), positive reinforcement (4-items), warmth (3-items), and supportiveness (3-items) sub-scales. Response options ranged from 1 (Never) to 5 (Always) reflecting the frequency with which parents engaged in different parenting behaviors.
Negative Parenting | Baseline, 2-month, and 4-month follow-up assessments.
  All parents completed the 18-item negative parenting composite measure of the Multidimensional Assessment of Parenting Scale, which was comprised of hostility (7-items), physical control (4-items), and lax control (7-items) sub-scales. Response options ranged from 1 (Never) to 5 (Always) reflecting the frequency with which parents engaged in different parenting behaviors.
Parental Psychological Control | Baseline, 2-month, and 4-month follow-up assessments.
  All parents completed the 8-item Parent Psychological Control Measure, that is based off the Psychological Control Scale - Youth Self-Report. Response options ranged from 1 (Never) to 5 (Always) reflecting the frequency with which parents engaged in different parenting behaviors.
Parental Knowledge of Effective Parenting Strategies | Baseline, 2-month, and 4-month follow-up assessments.
  All parents completed the 16-item Brief Version of the Knowledge of Parenting Strategies Scale. Parents selected one response that would reflect the most effective action for a parent to take in a situation described in the question.
Parental Hope | Baseline, weekly, through intervention completion (average of 3 weeks), 2-month, and 4-month follow-up assessments.
  All parents completed the 5-item Hope for Parenting Scale. Response options ranged from 1 (Definitely False) to 8 (Definitely True) indicating how much they agree or disagree with each item.
Parental Self-Efficacy | Baseline, weekly, through intervention completion (average of 3 weeks), 2-month, and 4-month follow-up assessments.
  All parents completed the 5-item Brief Parental Self-Efficacy Scale. Response options ranged from 1 (Strongly Disagree) to 5 (Strongly Agree), indicating how much they agreed with each statement.
Global Satisfaction | 2-months
  Parents assigned to an intervention condition also completed the 8-item Client Satisfaction Questionnaire. Response options ranged from 1 (None of my needs have been met, Quite dissatisfied) to 4 (Almost all of my needs have been met, Very satisfied).

SECONDARY OUTCOMES:
Child Emotional and Behavioral Difficulties | Baseline, 2-month, and 4-month follow-up assessments.
  All parents completed the 25-item Strengths and Difficulties Questionnaire. This measure consists of emotional problems (5-items), conduct problems (5-items), hyperactivity (5-items), peer problems (5-items), and prosocial behavior (5-items) sub-scales. Each sub-scale will be examined as an outcome, along with the total difficulties scale, which is a composite of all five sub-scales and reflects overall emotional and behavioral difficulties. Response options ranged from 0 (Not true) to 2 (Certainly True) and reflects how often children experience various difficulties.
Child Emotion Dysregulation | Baseline, 2-month, and 4-month follow-up assessments.
  All parents completed the 24-item Emotion Dysregulation Inventory. Response options ranged from 0 (Not at all) to 4 (Very severe) reflecting the severity of various emotions and behaviors displayed by children.
Child Emotion Regulation | Baseline, 2-month, and 4-month follow-up assessments.
  All parents completed the 8-item emotion regulation sub-scale of the Emotion Regulation Checklist. Response options ranged from 0 (Never) to 3 (Almost always) reflecting the frequency with which children displayed various emotions and behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: John L. Cooley, Ph.D., Principal Investigator — University of Florida
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sumargi A, Sofronoff K, Morawska A. A Randomized-Controlled Trial of the Triple P-Positive Parenting Program Seminar Series with Indonesian Parents. Child Psychiatry Hum Dev. 2015 Oct;46(5):749-61. doi: 10.1007/s10578-014-0517-8. PMID 25335876
- [Background] Sanders, M., Prior, J., & Ralph, A. (2009). An evaluation of a brief universal seminar series on positive parenting: A feasibility study. Journal of Children's Services, 4(1), 4-20. https://doi.org/10.1108/17466660200900002
- [Background] Foskolos, K., Gardner, F., & Montgomery, P. (2023). Brief parenting seminars for preventing child behavioral and emotional difficulties: A pilot randomized controlled trial. Journal of Child and Family Studies, 32(10), 3063-3075. https://doi.org/10.1007/s10826-023-02653-6